CLINICAL TRIAL: NCT07311551
Title: A Comparison of Effectiveness, Safety, and Cost-effectiveness of Dapagliflozin and Empagliflozin in Patients With Type 2 Diabetes Mellitus and High Body Mass Index (BMI): A Randomized Controlled Trial at a Tertiary Care Hospital in Central India
Brief Title: A Comparison of Effectiveness, Safety, and Cost-effectiveness of Dapagliflozin and Empagliflozin in Patients With Type 2 Diabetes Mellitus and High Body Mass Index (BMI)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bhavya Bhavya, MD (Other)
Responsible Party: Sponsor-Investigator, Bhavya Bhavya, MD, SENIOR RESIDENT, All India Institute of Medical Sciences
Organization: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ihecsr/aiimsbpl/July25/213
Record Dates: First submitted 2025-11-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes mellitus, MASLD, Overweight, Glycaemic effectivness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — dapagliflozin; Tablets; empagliflozin

STUDY DESIGN:
Intervention Model Description: This will be a prospective, randomized, open-label, parallel-group single-centre clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Dapagliflozin 10 mg given once daily per orally for 6 months
  Interventions: Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy
- Group B (Experimental): Empagliflozin 25mg given once daily per orally for 6 months
  Interventions: Drug: Empagliflozin (25 Mg Tab) along with standard medical therapy

INTERVENTIONS:
Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy — Group A: Dapagliflozin 10 mg once daily + Metformin ± OHAs
  Arms: Group A
Drug: Empagliflozin (25 Mg Tab) along with standard medical therapy — Group B: Empagliflozin 25 mg once daily + Metformin ± OHAs
  Arms: Group B

SUMMARY:
This study aims to compare the effect of two drugs used to treat diabetes, that is, Dapagliflozin and Empagliflozin on HbA1c (which is an indicator of blood sugar over the last 3 months) body weight, liver and kidney function, blood pressure, and overall cost-effectiveness in patients with type 2 diabetes and high body mass index (23kg/m2). The results will help us determine which drug is more effective, safer, and economical for Indian patients and improve future treatment options.

DETAILED DESCRIPTION:
The convergence of India's diabetes epidemic, high rates of obesity and MASLD, and the availability of pleiotropic SGLT2 inhibitors presents both an opportunity and a challenge for optimal diabetes management. While both dapagliflozin and empagliflozin provide significant benefits over and above glycemic control, the absence of direct comparative data in Indian populations limits evidence-based treatment decisions. This study aims to address these critical knowledge gaps by delivering comprehensive comparative effectiveness and cost-effectiveness data to inform clinical practice and healthcare policy in India.

Despite extensive evidence supporting the use of SGLT2 inhibitors, several important knowledge gaps remain, especially in relation to Indian clinical practice.

* Lack of head-to-head comparative data: No Indian randomized controlled trial has directly compared dapagliflozin and empagliflozin in terms of efficacy and safety in patients with type 2 diabetes mellitus (T2DM) and high body mass index.
* Limited data on hepatic outcomes: While individual studies indicate liver benefits, no research has systematically compared the two agents using established hepatic assessment methods such as controlled attenuation parameter (CAP) and liver stiffness measurement (LSM) via transient elastography.
* Population-specific considerations: Indian patients may respond differently to SGLT2 inhibitors due to genetic polymorphisms affecting drug metabolism, distinct body composition patterns, and diverse dietary and lifestyle influences.
* Economic evaluation gaps: There is a lack of comprehensive pharmacoeconomic analyses comparing these agents within the Indian healthcare system, which limits evidence-based formulary choices and reimbursement decisions.
* Real-world effectiveness: While efficacy is proven in controlled trial settings, data on real-world effectiveness in Indian clinical practice conditions remain limited.

This study is uniquely positioned to address this gap by conducting a head-to-head, RCT of dapagliflozin vs. empagliflozin in Indian adults with T2DM and high BMI. The design ensures standardized background therapy, minimizes bias, and includes a comprehensive evaluation of metabolic (HbA1c, weight), hepatic (CAP and LSM), renal, and cardiovascular outcomes, as well as adverse events and patient-reported tolerability. Furthermore, it incorporates a pharmacoeconomic analysis using Average and Incremental Cost-Effectiveness Ratios (ACER, ICER) to assess affordability and value, a key consideration in India and other low- and middle-income countries (LMICs).

By generating robust, context-specific data on comparative efficacy and value of these agents, this study aims to fill a crucial knowledge gap and support personalized clinical decision-making. It is thus expected to make a meaningful contribution to optimizing diabetes care in India.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older with a diagnosis of type 2 diabetes mellitus (T2DM) who have been on stable background therapy for at least three months were eligible for inclusion. Participants were required to have an HbA1c level between 7% and 10% while receiving Metformin with or without other oral hypoglycemic agents, and there had to be a clear clinical indication to initiate an SGLT2 inhibitor. Individuals with a body mass index (BMI) of 23 kg/m² or higher and who were willing to provide written informed consent were included in the study.

Exclusion Criteria:

Patients were excluded if they had uncontrolled diabetes with an HbA1c level greater than 10.0% or if they had used SGLT2 inhibitors, insulin, or GLP-1 receptor agonists within 90 days prior to randomization. Individuals with a history of bariatric surgery or those planning such surgery during the study period were not eligible. Current alcohol consumption of ≥140 g/week in women or ≥210 g/week in men-equivalent to at least 14 or 21 standard drinks per week, respectively-was also an exclusion criterion. Acutely ill patients visiting the OPD, those receiving medications known to cause hepatic steatosis (such as amiodarone, valproate, tamoxifen, methotrexate, or steroids), and individuals with an eGFR <45 mL/min/1.73 m² were excluded. Patients with contraindications to SGLT2 inhibitor use, including a history of recurrent urinary or genital infections, current or previous gangrene, known hypersensitivity to the drug, or a history of diabetic ketoacidosis, were also not included. Pregnant or breastfeeding women were excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-12-24 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from baseline at 6 months | From enrollment to the end of treatment at 6 months
Change in weight from baseline at 6 months | From enrollment to the end of treatment at 6 months

SECONDARY OUTCOMES:
Change in HbA1c (%) from baseline at 3 months | From enrollment to the end of treatment at 3 months
Change in FBG (mg/dL) from baseline at 6 months | From enrollment to the end of treatment at 6 months
Change in ALT from baseline at 6 months | From enrollment to the end of treatment at 6 months
Changes in LSM from baseline at 6 months | From enrollment to the end of treatment at 6 months
Change in SBP (mmHg) from baseline at 6 months | From enrollment to the end of treatment at 6 months
Change in serum creatinine (mg/dL) from baseline at 6 months | From enrollment to the end of treatment at 6 months
Incidence of adverse events from baseline at 6 month | From enrollment to the end of treatment at 6 months
Incidence of Drug-related Discontinuation at 6 month | From enrollment to the end of treatment at 6 months
Change in AST from baseline at 6 months | From enrollment to the end of treatment at 6 months
Changes in CAP from baseline at 6 months | From enrollment to the end of treatment at 6 months
Change in GGT from baseline at 6 months | From enrollment to 6 months
Change in DBP (mmHg) from baseline at 6 months | From enrollment to end of treatment at 6 months
Change in eGFR from baseline at 6 months | From enrollment to end of treatment at 6 months
Change in UACR (mg/g) from baseline at 6 months | From enrollment to end of treatment at 6 months

IPD SHARING:
Plan to Share IPD: Undecided